CLINICAL TRIAL: NCT00008346
Title: Screening and Diagnostic Trial to Compare the Effectiveness of Two Types of Mammography in Detecting Breast Cancer in Women
Brief Title: Digital Mammography Screening Trial (ACRIN6652)
Acronym: DMIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CDR0000068399; ACRIN-6652 (Other: American College of Radiology); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

ARMS (2):
- SFM then FFDM (Other): Screen Film Mammography (SFM) followed by Full Field Digital Mammography (FFDM)
  Interventions: Diagnostic Test: Full Field Digital Mammography; Diagnostic Test: Screen Film Mammography
- FFDM then SFM (Other): Full Field Digital Mammography (FFDM) followed by Screen Film Mammography (SFM)
  Interventions: Diagnostic Test: Full Field Digital Mammography; Diagnostic Test: Screen Film Mammography

INTERVENTIONS:
Diagnostic Test: Full Field Digital Mammography — Radiologic test to screen women for Breast cancer using digital detectors
  Other Names: FFDM; Digital Mammography
Diagnostic Test: Screen Film Mammography — Radiologic test to screen women for Breast cancer using plain film detectors a resolution screen
  Other Names: SFM; Plain Film Mamography

SUMMARY:
RATIONALE: Screening tests may help doctors detect cancer cells early and plan more effective treatment for cancer. It is not yet known which type of mammography is more effective in detecting breast cancer.

PURPOSE: Screening and diagnostic trial to compare the effectiveness of two types of mammography in detecting breast cancer in women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the diagnostic performance of digital mammography vs screen-film mammography, as measured by the area under the Receiver Operating Characteristic (ROC) curve, sensitivity, specificity, and positive and negative predictive values, in the detection of breast cancer in women.
* Compare the diagnostic accuracy of the digital mammogram obtained using each of the individual manufacturer's digital units vs screen-film mammography through retrospective reader studies.
* Determine the effects of patient characteristics, including age, lesion type, pathologic diagnosis, menopausal and hormonal status, breast density, and family history, on diagnostic accuracy of digital mammography.
* Determine the effects of technical parameters, including display type, machine type, and detector spatial and contrast resolution, on diagnostic accuracy of digital mammography.
* Determine the effect of reduced false-positive mammograms that are expected with digital mammography on the health-related quality of life and personal anxiety of women undergoing this screening experience.
* Compare the diagnostic performance of digital mammography with the rate of cancer in a set of cases through a retrospective reader study.
* Compare the effect of softcopy vs printed film display on the diagnostic performance of digital mammography through a retrospective reader study.
* Compare the effect of breast density on the diagnostic accuracy of digital mammography vs screen-film mammography through a retrospective reader study.
* Compare the image quality and breast radiation dose in digital vs screen-film mammography in these participants.
* Determine the temporal variations in image quality, breast radiation dose, and other quality control parameters in the participating study centers.

OUTLINE: This is a randomized, multicenter study. Participants with postitive screening results are stratified according to age (under 50 vs 50-59 vs 60-70 vs over 70). Participants are randomized to one of two treatment arms.

* Arm I: Participants undergo a two-view screen-film mammogram followed by a two-view digital mammogram of each breast.
* Arm II: Participants undergo a two-view digital mammogram followed by a two-view screen-film mammogram of each breast.

Quality of life is assessed before the screening mammogram in the first 800 women enrolled. In an additional 1,200 participants (600 with positive screening results and 600 with negative screening results), quality of life is assessed shortly after the screening mammogram and at 1 year.

Participants are followed at 1 year with a repeat screen-film or digital mammogram.

PROJECTED ACCRUAL: A total of 49,500 participants (24,750 per arm) will be accrued for this study within 18 months.

ELIGIBILITY:
4.1 Inclusion Criteria 4.1.1 All consecutive women presenting for screening mammography at the participating institutions will be eligible.

4.1.2 Signed study-specific informed consent. See Appendix I. 4.2 Exclusion Criteria 4.2.1 All women who have presented with a complaint of a focal dominant lump or a bloody or clear nipple discharge.

4.2.2 All women who have breast implants. 4.2.3 Any woman who is pregnant or has reason to believe that she might be pregnant.

4.2.4 Participants who cannot, for any reason, undergo follow-up screen-film mammography at the participating institution or provide mammograms from another institution for review for one year after study entry.

4.2.5 All women with a history of breast cancer treated with lumpectomy. Note: Women with a history of breast cancer treated with mastectomy who have now returned to a screening population will still be included in the study.

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49528 (Actual)
Dates: Start 2001-10 (Actual); Primary Completion 2005-02 (Actual); Study Completion 2005-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etta Pisano, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (32):
- United States (31):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Washington Radiology Associates, P.C., Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory Health Care Clinic, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Shore Memorial Hospital, Somers Point, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Elizabeth Wende Breast Clinic, Rochester, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Sunnybrook and Women's College Health Sciences Centre, North York, Ontario, Canada

REFERENCES:
- [Background] Hendrick RE, Pisano ED, Averbukh A, Moran C, Berns EA, Yaffe MJ, Herman B, Acharyya S, Gatsonis C. Comparison of acquisition parameters and breast dose in digital mammography and screen-film mammography in the American College of Radiology Imaging Network digital mammographic imaging screening trial. AJR Am J Roentgenol. 2010 Feb;194(2):362-9. doi: 10.2214/AJR.08.2114. PMID 20093597
- [Background] Tosteson AN, Stout NK, Fryback DG, Acharyya S, Herman BA, Hannah LG, Pisano ED; DMIST Investigators. Cost-effectiveness of digital mammography breast cancer screening. Ann Intern Med. 2008 Jan 1;148(1):1-10. doi: 10.7326/0003-4819-148-1-200801010-00002. PMID 18166758
- [Result] Baum JK, Hanna LG, Acharyya S, Mahoney MC, Conant EF, Bassett LW, Pisano ED. Use of BI-RADS 3-probably benign category in the American College of Radiology Imaging Network Digital Mammographic Imaging Screening Trial. Radiology. 2011 Jul;260(1):61-7. doi: 10.1148/radiol.11101285. Epub 2011 Apr 18. PMID 21502382
- [Result] Hendrick RE, Cole EB, Pisano ED, Acharyya S, Marques H, Cohen MA, Jong RA, Mawdsley GE, Kanal KM, D'Orsi CJ, Rebner M, Gatsonis C. Accuracy of soft-copy digital mammography versus that of screen-film mammography according to digital manufacturer: ACRIN DMIST retrospective multireader study. Radiology. 2008 Apr;247(1):38-48. doi: 10.1148/radiol.2471070418. PMID 18372463
- [Result] Pisano ED, Hendrick RE, Yaffe MJ, Baum JK, Acharyya S, Cormack JB, Hanna LA, Conant EF, Fajardo LL, Bassett LW, D'Orsi CJ, Jong RA, Rebner M, Tosteson AN, Gatsonis CA; DMIST Investigators Group. Diagnostic accuracy of digital versus film mammography: exploratory analysis of selected population subgroups in DMIST. Radiology. 2008 Feb;246(2):376-83. doi: 10.1148/radiol.2461070200. PMID 18227537
- [Result] Bloomquist AK, Yaffe MJ, Pisano ED, Hendrick RE, Mawdsley GE, Bright S, Shen SZ, Mahesh M, Nickoloff EL, Fleischman RC, Williams MB, Maidment AD, Beideck DJ, Och J, Seibert JA. Quality control for digital mammography in the ACRIN DMIST trial: part I. Med Phys. 2006 Mar;33(3):719-36. doi: 10.1118/1.2163407. PMID 16878575
- [Result] Yaffe MJ, Bloomquist AK, Mawdsley GE, Pisano ED, Hendrick RE, Fajardo LL, Boone JM, Kanal K, Mahesh M, Fleischman RC, Och J, Williams MB, Beideck DJ, Maidment AD. Quality control for digital mammography: part II. Recommendations from the ACRIN DMIST trial. Med Phys. 2006 Mar;33(3):737-52. doi: 10.1118/1.2164067. PMID 16878576
- [Result] Pisano ED, Gatsonis CA, Yaffe MJ, Hendrick RE, Tosteson AN, Fryback DG, Bassett LW, Baum JK, Conant EF, Jong RA, Rebner M, D'Orsi CJ. American College of Radiology Imaging Network digital mammographic imaging screening trial: objectives and methodology. Radiology. 2005 Aug;236(2):404-12. doi: 10.1148/radiol.2362050440. Epub 2005 Jun 16. PMID 15961755
- [Result] Pisano ED, Gatsonis C, Hendrick E, Yaffe M, Baum JK, Acharyya S, Conant EF, Fajardo LL, Bassett L, D'Orsi C, Jong R, Rebner M; Digital Mammographic Imaging Screening Trial (DMIST) Investigators Group. Diagnostic performance of digital versus film mammography for breast-cancer screening. N Engl J Med. 2005 Oct 27;353(17):1773-83. doi: 10.1056/NEJMoa052911. Epub 2005 Sep 16. PMID 16169887